CLINICAL TRIAL: NCT03236974
Title: An Open Label, Randomised, Pre-surgical, Pharmacodynamics Study to Compare the Biological Effects of AZD9496 Versus Fulvestrant in Postmenopausal Women With ER Positive HER-2 Negative Primary Breast Cancer
Brief Title: Study to Compare the Effects of AZD9496 vs Fulvestrant in Breast Cancer.
Acronym: D6090C00002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6090C00002
Record Dates: First submitted 2017-07-18; First posted 2017-08-02 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Postmenopausal Women With ER+ HER2- Primary Breast Cancer
MeSH Terms: interventions — Fulvestrant; AZD9496; Drug Evaluation

STUDY DESIGN:
Masking Description: Not applicable, thisis an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (Active Comparator): Fulvestrant, 500 mg
  Interventions: Drug: Standard Arm - Fulvestrant
- AZD9496 (Experimental): 250 mg bd taken orally for 5-14 days
  Interventions: Drug: AZD9496

INTERVENTIONS:
Drug: Standard Arm - Fulvestrant — 500 mg Fulvestrant administered as two consecutive 5 ml intramuscular injections on Day 1, one in each buttock
  Other Names: Fulvestrant
  Arms: Standard arm
Drug: AZD9496 — Administered at 250 mg bd orally for 5-14 days commencing on Day 1, and continuing up to the day of biopsy
  Other Names: Study drug
  Arms: AZD9496

SUMMARY:
This is an open label randomised multicentre pre-surgical pharmacodynamics study to compare and assess the biological effects of AZD9496 and fulvestrant in postmenopausal women with estrogen receptor (ER) positive (ER+), human epidermal growth factor receptor 2 (HER-2) negative (HER2-) primary breast cancer.

Patients will receive AZD9496 or fulvestrant and will have an on-treatment image

-guided core biopsy after 5-14 days of commencing treatment.

DETAILED DESCRIPTION:
This is an open label, randomized, multi-centre study in postmenopausal women with primary ER+ HER2- breast cancer. Patients will be randomised to an oral dose of 250 mg bd AZD9496 or 500mg fulvestrant i.m. administered on one occasion. Patients diagnosed with primary breast cancer who are scheduled for surgery with curative intent will be consented to the study including consent to use the formalin fixed paraffin embedded (FFPE) diagnostic tumor biopsy sample and fresh frozen tumor biopsy sample (if available) for research purposes. Patients may also consent to provide an optional pretreatment fresh frozen tumor biopsy sample if this was not obtained at the time of initial diagnostic biopsy. If the diagnostic biopsy was taken ≥ 6 weeks prior to starting treatment or was not of sufficient quality, new tumor core biopsies (FFPE and fresh frozen) must be taken. Following the screening visit, eligible patients will be randomised to receive one of the following study treatments:

* AZD9496 administered at 250 mg bd orally for 5-14 days commencing on Day 1, and continuing up to the day of biopsy OR
* fulvestrant 500 mg administered as two consecutive 5 ml intramuscular injections on Day 1, one in each buttock.

After the morning dose of AZD9496 on the day of biopsy dosing will be stopped. If following initiation of AZD9496 treatment, dosing will be stopped if biopsy is postponed beyond Day 14. Patients will be considered not evaluable for the study if biopsy is postponed beyond day 14 of AZD9496/fulvestrant treatment initiation. Core tumor biopsies will be taken at either the time of definitive surgery or at a separate visit prior to surgery in the period between (and including) day 5 and day 14. Subjects who are scheduled to start a subsequent neoadjuvant therapy must have their core tumor biopsies performed before commencing neoadjuvant treatment.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated informed consent form (ICF)
2. Women >=18 years
3. Patients with newly diagnosed resectable primary breast cancer scheduled to undergo treatment with curative intent by surgery
4. Histologically confirmed invasive breast cancer involving a palpable tumor of any size, or a tumor with an ultrasound assessed diameter of ≥ 1.0 cm
5. Any clinical nodal status
6. ER+breast cancer
7. HER2- breast cancer defined as a negative in situ hybridization test or an immno-histochemistry (IHC) status of 0 or 1+
8. Eastern Co-operative Oncology group (ECOG) performance status 0-1
9. Post-menopausal status defined as meeting at least one of the following criteria: Have undergone a bilateral oophorectomy; Age ≥60 years; Age ≥50 years and with cessation of regular menses ≥12 months and with an intact uterus in the absence of oral contraception or hormone-replacement therapy (HRT) prior to the diagnosis of breast cancer; Age <60 years and with cessation of regular menses ≥12 months and follicle stimulating hormone (FSH) and oestradiol levels in the postmenopausal range

Exclusion criteria:

1. Pre-treatment biopsy sample not likely to provide adequate tissue sections for the biomarker assays
2. Previous systemic or local treatment for the new primary breast cancer currently under investigation (including surgery, radiotherapy, cytotoxic and endocrine treatments)
3. Inflammatory breast cancer
4. Evidence of metastases
5. Patients currently receiving medications or herbal supplements known to be strong inhibitors/inducers of CYP3A4/5 or strong inhibitors of CYP2C8 or that are sensitive substrates of CYP2C8 inhibition
6. Concurrent treatment with other experimental drugs within 4 weeks prior to receiving study treatment
7. Use of hormone-replacement therapy from <4 weeks of the diagnostic/baseline core biopsy to the start of trial treatment
8. Patients with second primary cancer. Any endocrine therapies or other anti-cancer therapies must have been ceased at least 12 months prior to enrollment.
9. Any of the following cardiac criteria:

   * Mean resting QT interval corrected for heart rate (QTc) > 470 msec obtained from 3 ECGs using Fridericia's formula
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
10. Experience of any of the following in the preceding 6 months: coronary artery bypass graft (CABG), angioplasty, vascular stent, myocardial infarction (MI), angina pectoris, congestive heart failure New York Heart Association (NYHA) Grade ≥2, cerebrovascular accident (CVA), transient ischaemic attack (TIA), deep venous or arterial thrombosis, pulmonary embolism, bleeding diathesis (i.e., disseminated intravascular coagulation, clotting factor deficiency) or requirement of anticoagulant therapy
11. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases,
12. Uncontrolled symptomatic thyroid dysfunction (hyperthyroidism or hypothyroidism).
13. Unexplained symptomatic endometrial disorders.
14. Refractory nausea and vomiting, uncontrolled chronic GI diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9496.
15. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: absolute neutrophil count < 1.5 x 109/L, Platelet count < 100 x 109/L, Haemoglobin < 90 g/L, alanine aminotransferase (ALT) > 2.5x upper limit of normal (ULN), aspartate aminotransferase (AST) > 2.5 x ULN, Total bilirubin > 1.5 x ULN or > 3 x in case of Gilbert's Syndrome, glomerular filtration rate < 50 mL/min
16. Direct involvement in the planning and conduct of the study
17. History of hypersensitivity to AZD9496
18. History of hypersensitivity to fulvestrant and/or castor oil
19. Judgment by the investigator that the patient should not participate in the study if unlikely to comply with study procedures, restrictions and requirements In addition, the following is considered a criterion for exclusion from the exploratory genetic research: Previous allogeneic bone marrow transplant; Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics changes to estrogen receptor (ER) expression following treatment with AZD9496 or fulvestrant | Tumour biopsy taken at baseline within 6 weeks of planned start of study treatment; on-treatment tumour biopsy taken following 5-14 day on study treatment
  Evaluation of AZD9496 and fulvestrant activity in the tumour by assessment of pharmacodynamics biomarker changes i.e. ER expression

SECONDARY OUTCOMES:
Pharmacodynamics changes to progesterone receptor (PgR) expression following treatment with AZD9496 or fulvestrant | Tumour biopsy taken at baseline within 6 weeks of planned start of study treatment; on-treatment tumour biopsy taken following 5-14 day on study treatment
  Evaluation of AZD9496 and fulvestrant activity in the tumour by assessment of pharmacodynamics biomarker changes i.e. PgR expression
Pharmacodynamics changes to Ki67 protein biomarker expression following treatment with AZD9496 or fulvestrant | Tumour biopsy taken at baseline within 6 weeks of planned start of study treatment; on-treatment tumour biopsy taken following 5-14 day on study treatment
  Evaluation of AZD9496 and fulvestrant activity in the tumour by assessment of pharmacodynamics biomarker changes i.e. Ki67 protein biomarker expression
Safety and tolerability of AZD9496 | From first dose until 28 days after last dose of AZD9496
  Safety and tolerability will be assessed in terms of adverse events (AEs), laboratory data, vital signs and ECG changes.
Safety and tolerability of fulvestrant | From first dose until 28 days after fulvestrant
  Safety and tolerability will be assessed in terms of adverse events (AEs), laboratory data and vital signs
Plasma concentration of AZD9496 - stand alone biopsy visit option | Blood samples collected close as possible to time of biopsy, 1-2 hours after biopsy and optional 3-4 hours after biopsy
  Determination of AZD9496 concentrations in plasma
Plasma concentration of fulvestrant | A blood sample will be collected anytime before biopsy.
  Determination of fulvestrant concentration in plasma
Plasma concentration of AZD9496 - on the table biopsy option | Blood samples collected close as possible to time of biopsy, at least 2 hours after biopsy and 8-12 hours after last dose or at discharge which is defined as up to 12 hours after last dose
  Determination of AZD9496 concentration in plasma

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (4):
  - Research Site, Erlangen
  - Research Site, Minden
  - Research Site, München
  - Research Site, Schwerin
- United Kingdom (6):
  - Research Site, Derby
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Poole
  - Research Site, Sutton in Ashfield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Robertson JFR, Evans A, Henschen S, Kirwan CC, Jahan A, Kenny LM, Dixon JM, Schmid P, Kothari A, Mohamed O, Fasching PA, Cheung KL, Wuerstlein R, Carroll D, Klinowska T, Lindemann JPO, MacDonald A, Mather R, Maudsley R, Moschetta M, Nikolaou M, Roudier MP, Sarvotham T, Schiavon G, Zhou D, Zhou L, Harbeck N. A Randomized, Open-label, Presurgical, Window-of-Opportunity Study Comparing the Pharmacodynamic Effects of the Novel Oral SERD AZD9496 with Fulvestrant in Patients with Newly Diagnosed ER+ HER2- Primary Breast Cancer. Clin Cancer Res. 2020 Aug 15;26(16):4242-4249. doi: 10.1158/1078-0432.CCR-19-3387. Epub 2020 Mar 31. PMID 32234755
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Search